CLINICAL TRIAL: NCT05410249
Title: Assessment of FOXP3 Gene Polymorphisms and Serum Interleukin 10 and Their Clinical Significance in Adult Patients With Immune Thrombocytopenia
Brief Title: Assessment of FOXP3 Gene Polymorphisms and Serum Interleukin 10 in Patients With ITP
Acronym: FoxP3ITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer of medical microbiology and immunology, faculty of medicine, Sohag University
Other Study IDs: Soh-Med-22-4-34
Record Dates: First submitted 2022-05-27; First posted 2022-06-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Thrombocytopenia
Keywords: polymorphism; FOXp3; serum IL10
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — !0 ml blood will be aspirated from the both groups and will be subjected to the following investigations:
  1. Complete blood count.
  2. Renal and liver function tests.
  3. Serology for HCV, HBV, and HIV.
  4. Antinuclear antibody
  5. Bone marrow examination.
  6. Serum IL-10 by enzyme-linked immunosorbent assay (ELISA).
  7. Genotyping of -6054 del/ATT and -924 A/G polymorphisms was performed using the real-time polymerase chain reaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primary ITP: Patients with primary ITP and aged 18 and older will be included in the study. Patients under 18 and those with proven secondary ITP [as cases initiated by or associated with infections due to human immunodeficiency virus (HIV-associated), hepatitis B virus, or hepatitis C virus-associated secondary ITP] will be excluded. Moreover, patients with accompanying autoimmune disorders such as systemic lupus erythematosus (SLE) and patients of malignancies were excluded.
  Interventions: Diagnostic Test: Serum IL10 By ELISA; Diagnostic Test: SNP -3279 A/C of FOXP3; Diagnostic Test: SNP-924 A/G Of FOXP3
- normal individuals: The control group will be age-matched and sex-matched normal healthy volunteers.
  Interventions: Diagnostic Test: Serum IL10 By ELISA; Diagnostic Test: SNP -3279 A/C of FOXP3; Diagnostic Test: SNP-924 A/G Of FOXP3

INTERVENTIONS:
Diagnostic Test: Serum IL10 By ELISA — measurement Of IL10 by ELISA
Diagnostic Test: SNP -3279 A/C of FOXP3 — Genotyping of -6054 del/ATT will be performed using the real-time polymerase chain reaction.
Diagnostic Test: SNP-924 A/G Of FOXP3 — Genotyping of -924 A/G polymorphisms was performed using the real-time polymerase chain reaction.

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune condition characterized by increased platelet destruction and suppression of production resulting in isolated thrombocytopenia. The exact etiology of ITP is unknown; however, multiple disease mechanisms exist and are mostly related to immune dysregulation [1].

Many studies in recent years have indicated that regulatory T cells (Tregs) play a critical role in the maintenance of immunological tolerance, and they have been reported to be defective in ITP patients, either numerically or functionally. [2-6]. They inhibit the activation and proliferation of effector T cells by the secretion of cytokines such as interleukin-10 (IL-10) and tumor growth factor-β (TGF-β) and by cell-to-cell interaction [7, 8].

DETAILED DESCRIPTION:
The suppressor function of Treg cells may be compromised if the FOXP3 gene is deficient. FOXP3 gene single nucleotide polymorphisms (SNPs), particularly regulatory polymorphisms in the promoter regions, have been linked to a variety of autoimmune diseases, including allergic rhinitis, type I diabetes (TID), systemic lupus erythematosus (SLE), multiple sclerosis (MS), and autoimmune thyroid diseases (AITD), according to numerous studies [9-13].

The FOXP3 gene's promoter region, which is crucial in gene expression and Treg activation, may contain important SNPs. The 6054 del/ATT and 924A > G SNPs are functionally well-defined and are distinguished by the relevance of studies on them among these SNPs. [14, 15].

The Interleukin 10 (IL-10) cytokine is required for regulating immune functions by promoting the widespread suppression of immune responses through its pleiotropic effects. IL-10 secretion from CD4+CD25+FoxP3+ regulatory cells (Tregs), macrophages and other leukocytes followed by subsequent binding to IL-10 receptors on macrophages and dendritic cells (DCs) has been linked to reduced antigen presentation and increased T-cell anergy [16]. The relationship between the two FOXP3 polymorphisms and ITP has not been well elucidated, hence the objective of this study is to explore if these functional polymorphisms are linked to ITP, how they correlate to IL-10 levels, and how they relate to other features of clinical presentation in adult patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary ITP and aged 18 and older will be included in the study.

Exclusion Criteria:

1. Patients under 18 and those with proven secondary ITP [as cases initiated by or associated with infections due to human immunodeficiency virus (HIV-associated), hepatitis B virus, or hepatitis C virus-associated secondary ITP] .
2. Patients with accompanying autoimmune disorders such as systemic lupus erythematosus (SLE).
3. Patients with malignancies will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary ITP and aged 18 and older will be included in the study. Patients under 18 and those with proven secondary ITP [as cases initiated by or associated with infections due to human immunodeficiency virus (HIV-associated), hepatitis B virus, or hepatitis C virus-associated secondary ITP] will be excluded. Moreover, patients with accompanying autoimmune disorders such as systemic lupus erythematosus (SLE) and patients of malignancies were excluded.
  All patients will be subjected to a thorough assessment of history, complete clinical examination, and investigations
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
SNP effect in FOXP3 gene in patients ITP | 26 May to August 2022
  different genotypes of FOXP3 in patients with ITP will be determined using real time PCR
Association of serum IL-10 levels in both groups( patients with ITP and normal control) | 26 May to August 2022
  measurement of serum IL10 in patients with ITP and normal controls using ELISA
Association of SNP in FOXP3 gene and the clinical presentation in adult patients with ITP | 26 May to August 2022
  evaluation and statistical analysis of effect of SNP in FOXP3 in the clinical picture in adult patients with ITP

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A Abdelbaset, lecturer, Principal Investigator — faculty of medicine, Sohag university
Locations (1):
- Faculty Of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballantine LE, Ong J, Midgley A, Watson L, Flanagan BF, Beresford MW. The pro-inflammatory potential of T cells in juvenile-onset systemic lupus erythematosus. Pediatr Rheumatol Online J. 2014 Jan 16;12:4. doi: 10.1186/1546-0096-12-4. PMID 24433387